CLINICAL TRIAL: NCT01052246
Title: The Pulsed Dye Laser as an Adjuvant Treatment Modality in Acne Vulgaris - a Randomized Controlled Single Blinded Trial
Brief Title: Pulsed Dye Laser Treatment of Acne Vulgaris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laserklinik Karlsruhe (Other)
Responsible Party: Syrus Karsai/Principal investigator, Laserklinik Karlsruhe
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LK_08_2009
Record Dates: First submitted 2010-01-19; First posted 2010-01-20 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Acne Vulgaris
Keywords: acne vulgaris; laser surgery; pulsed dye lasers; benzoyl peroxidase; clindamycin; randomized controlled trial
MeSH Terms: conditions — Acne Vulgaris | interventions — Lasers, Dye

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clindamycin 1% + benzoyl peroxide 5% & pulsed dye laser (Experimental)
  Interventions: Device: Pulsed dye laser
- Clindamycin 1% + benzoyl peroxide 5% (Active Comparator)
  Interventions: Drug: Fixed combination of clindamycin 1% + benzoyl peroxide 5%

INTERVENTIONS:
Drug: Fixed combination of clindamycin 1% + benzoyl peroxide 5% — Topical monotherapy with a fixed combination of 1% clindamycin and 5% benzoyl peroxide hydrating gel (Duac® Akne Gel, Stiefel Laboratorium GmbH, Offenbach, Germany). In order to provide standardized condition within the sample, the gel was applied on the whole face regardless of the lesion location. The gel was applied once per day in the evening throughout the observation period and left in place overnight.
  Arms: Clindamycin 1% + benzoyl peroxide 5%
Device: Pulsed dye laser — Patients randomized in the experimental group received two additional treatments with a pulsed dye laser using the following parameters:
  * Wavelength 585 nm
  * Energy fluence 3 J/cm2
  * Pulse duration 0.35 msec
  * Spot size 7 mm
  Arms: Clindamycin 1% + benzoyl peroxide 5% & pulsed dye laser

SUMMARY:
The results of pulsed dye laser (PDL) treatment of acne vulgaris published so far are controversial: Whereas Seaton et al. described a marked improvement of mild-to-moderate acne after low-fluence pulsed-dye laser therapy, Orringer et al. were unable to replicate said results in a similar, albeit not identical, study design. More recently published studies failed to resolve the controversy, varying in terms of treatment procedure(s) as well as results.

While published results are certainly promising enough to be followed up by independent research, they are insufficient to justify the abdication of methods with proven efficacy. Considering patient treatment ethics and the short 'window of opportunity' for scar prevention when active inflammatory lesions are present, the investigators planned the adjuvant application of the PDL in the present study, providing all patients with the well established and evidentially effective modality of a fixed-combination clindamycin 1%-benzoyl peroxide 5% hydrating gel (C/BPO). The goal of the study was the assessment of the efficacy and safety of a low-fluence PDL treatment in addition to C/BPO in patients with facial inflammatory acne.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents and adults with moderate inflammatory acne vulgaris (ISGA degrees 2-4)
* Fitzpatrick skin type I-III

Exclusion Criteria:

* Atopic dermatitis
* Oral antibiotics during the last 4 weeks prior to enrolment
* Oral isotretinoin during the last 52 weeks prior to enrolment
* Oral contraceptives during the last 26 weeks prior to enrolment
* Topical acne therapeutics during the last 4 weeks prior to enrolment
* Diagnosis or anamnestic indication of a regional enteritis, Morbus Crohn or antibiotics-associated colitis
* Laser surgery interventions within the treatment region during the last 12 weeks prior to enrolment
* Coagulation anomalies or anticoagulant treatment
* Photo-sensitizing medication (e. g., tetracycline, gold)
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Investigator's Static Global Assessment | day 0, day 14, day 28
Lesions count | day 0, day 28

SECONDARY OUTCOMES:
Dermatology Life Quality Index | day 0, day 28
Documentation of side effects | day 28

CONTACTS AND LOCATIONS:
Overall Officials: Syrus Karsai, MD, Principal Investigator — Laserklinik Karlsruhe
Locations (1):
- Laserklinik Karlsruhe, Karlsruhe, Germany